CLINICAL TRIAL: NCT03880422
Title: Nutrition and Exercise Interventions to Reduce Androgen Deprivation Therapy-Induced Obese Frailty in Survivors of Advanced Prostate Cancer
Brief Title: Nutrition and Exercise Interventions in Reducing Androgen Deprivation Therapy-Induced Obese Frailty in Prostate Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 72118; NCI-2019-00341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 72118 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-03-01; First posted 2019-03-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cancer Survivor; Obesity; Overweight; Prostate Adenocarcinoma; Stage A Prostate Cancer; Stage B Prostate Cancer; Stage C Prostate Cancer; Stage D Prostate Cancer; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage IIC Prostate Cancer; Stage III Prostate Cancer; Stage IIIA Prostate Cancer; Stage IIIB Prostate Cancer; Stage IIIC Prostate Cancer; Stage IV Prostate Cancer; Stage IVA Prostate Cancer; Stage IVB Prostate Cancer
MeSH Terms: conditions — Obesity; Overweight; Prostatic Neoplasms | interventions — Diet Therapy; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (diet, exercise, education) (Experimental): Patients receive an individualized diet plan for 6 months. Patients complete an individualized home-based exercise program aerobic and resistance exercise over 10-30 minutes per day, at minimum 3 days per week for 6 months, and a progressive resistance exercise program including an individually tailored prescription targeting the chest, shoulders, arms, and leg musculature for 1-4 sets of 10-15 repetitions, 5 days per week over 6 months. Patients also attend monthly educational meetings for 6 months.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Educational Intervention; Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Receive diet plan
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Educational Intervention — Attend educational meeting
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Exercise Intervention — Complete exercise program
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies how well nutrition and exercise interventions work in reducing androgen deprivation therapy-induced obese frailty in prostate cancer survivors. Individualized nutrition and exercise advice for prostate cancer patients on androgen deprivation therapy may help to reduce obese frailty and change the levels of myokines in blood.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the effect of individualized nutrition and exercise counseling interventions on myokine expression and body composition in prostate cancer (PrCa) patients being treated with androgen deprivation therapy (ADT).

SECONDARY OBJECTIVES:

I. Determine any changes in muscle strength, respiratory muscle strength and functional capacity resulting from the nutrition and exercise counseling interventions.

II. Determine any changes in myokines, circulating inflammatory and frailty-associated cytokines resulting from the nutrition and exercise counseling interventions.

III. Determine the effect of the study interventions on dietary intake, physical activity, fatigue, and quality of life.

EXPLORATORY OBJECTIVES:

I. Correlate changes in secondary objectives with prostate specific antigen (PSA) and testosterone levels.

II. Evaluate adherence to nutrition and exercise advice. III. Evaluate assessment tools and recruiting strategies.

OUTLINE:

Patients receive an individualized diet plan for 6 months. Patients complete an individualized home-based exercise program aerobic and resistance exercise over 10-30 minutes per day, at minimum 3 days per week for 6 months, and a progressive resistance exercise program including an individually tailored prescription targeting the chest, shoulders, arms, and leg musculature for 1-4 sets of 10-15 repetitions, 5 days per week over 6 months. Patients also attend monthly educational meetings for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed prostate adenocarcinoma of any stage/grade
* Prescribed or already receiving continuous ADT for < 5 years
* Hemoglobin > 11 g/dL
* Creatinine < 1.5 x upper limit of normal (ULN), AST or ALT <2 x ULN within 6 months prior to enrollment
* Liver function tests < 2 x ULN
* Able to walk unassisted at least 100 meters (200 steps) or ECOG <= 1
* No contraindications to any aspect of participation, including aerobic exercise
* Participant must be able to read, write, and understand the English language and be able to provide written consent
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Known clinically significant severe chronic obstructive pulmonary disease (COPD), ischemic heart disease, congestive heart failure, and/or significant cardiac arrhythmias
* Limiting orthopedic, musculoskeletal or psychological conditions (clinician discretion)
* Overall medical frailty (clinician discretion)
* Any condition contraindicating additional blood collection beyond standard of care
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2029-05-02 (Estimated); Study Completion 2029-05-02 (Estimated)

PRIMARY OUTCOMES:
Changes in body composition | Baseline up to 6 months
  Will be measured by dual X-ray absorptiometry (DXA) total body and regional lean mass, fat mass and % body fat.

SECONDARY OUTCOMES:
Changes in muscle strength | Baseline up to 6 months
  Will be assessed by chest press, leg press, grip strength,6-minute walk test, timed-up-and-go, agility, Berg balance scale, short physical performance battery (SPPB).
Changes in functional capacity muscle strength | Baseline up to 6 months
  Improvement of muscle strenght
Change in body composition | Baseline up to 6 months
  All subjects will undergo dual-energy X-ray absorptiometry (DEXA) for measurements of body composition
myokines concentration | Baseline up to 6 months
  Will be assessed by serum biomarker levels.
cytokines concentration | Baseline up to 6 months
  Will be assessed by serum biomarker levels.
Health related quality of life Short Form | Up to 6 months
  Will be used to assess quality of life . The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100, Lower scores = more disability, higher scores = less disability
Changes in dietary intake | Baseline up to 6 months
  Will be assessed by National Cancer Institute Automated Self-Administered 24-hour survey.
Changes in physical activity | Baseline up to 6 months
  Will be assessed by Godin Leisure Time survey and Fitbit activity report. Will be summarized by time point using the observed sample size, mean, and standard deviation. Will be evaluated using a two-sided permutation paired t-test. Additionally, the mean change in each outcome will be estimated using a 95% confidence interval. As exploratory analyses, the association between the change in each outcome and demographic/clinical factors may be evaluated using general linear models. The change in outcome will be modeled as a function of baseline levels and each demographic/clinical factor in a one-at-a-time manner.
Change in fatigue | Baseline up to 6 months
  Will be assessed by the Functional Assessment of Chronic Illness Therapy-Fatigue survey.
Change in Respiratory Muscle Strength | Baseline up to 6 months
  Mouth pressure device

OTHER OUTCOMES:
Serum prostate specific antigen (PSA) and androgen levels | Up to 6 months
  Will evaluate the association between changes in the primary biomarkers with serum PSA and androgen levels.
Adherence to nutrition and exercise advice | Up to 6 months
  Adherence to advice is qualitative in nature and will be summarized using the appropriate descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal S Chatta, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States